CLINICAL TRIAL: NCT01958736
Title: Ballistic Strength Training in Stroke: A Phase II Randomized, Controlled, Assessor Blinded Pilot Study
Brief Title: Ballistic Strength Training in Stroke: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Australian Catholic University (Other)
Responsible Party: Principal Investigator, Ms. Rowan Frew, Ms. Rowan Frew, Bayside Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 369/13
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Ballistic Strength Training
  Interventions: Other: Ballistic Strength Training
- Control (Active Comparator): Usual care Physiotherapy
  Interventions: Other: Usual Care Physiotherapy

INTERVENTIONS:
Other: Ballistic Strength Training — The experimental group will complete jump squats on the leg sled, single leg toe push offs (or bilateral where unable to complete single), alternating legs (i.e. bounding), mini tramp jumping, progressing to jogging, quick hip flexion and bounding on land.
  Arms: Experimental
Other: Usual Care Physiotherapy — This group will complete a suite of exercises based upon existing rehabilitation practices that aim to improve mobility after stroke. The supervising physiotherapist will select and progress the exercises, recording the performance of exercises in an exercise log and detailing incidence of adverse events. Exercise selection will include: gait retraining, cardiovascular fitness, lower limb strengthening, static and dynamic balance.
  Arms: Control

SUMMARY:
This pilot study intends to evaluate whether stroke patients can complete ballistic strength exercises for thirty minutes, three times per week over a six week training period in addition to their existing rehabilitation program.

It will evaluate whether using ballistic training principles, is superior in improving mobility compared with usual care exercises to improve mobility and leg strength in stroke patients.

In this study there will be 15 participants per group, a total of 30 participants. The control group will receive usual care consistent with existing rehabilitation practice and literature. The experimental group will perform task specific strength training in a ballistic fashion.

DETAILED DESCRIPTION:
Research Aims:

1. To establish the feasibility of ballistic strength training in stroke and
2. To evaluate the effects of ballistic strength training exercises on mobility outcomes, strength and quality of life when compared with usual care.

Methods:

This wil be a prospective, randomized, controlled, assessor-blinded pilot study. It will be conducted 3 x per week for 6 weeks (i.e. a total of 18 sessions lasting 30 minutes).

Primary outcome measure: Feasibility

* Recruitment
* Retention/Attrition
* Clinical Feasibility
* Safety

Secondary outcome measures - measured at baseline and completion

* Ten metre walk test (10MWT) comfortable pace
* 10MWT maximum safe pace
* High level mobility assessment tool (HiMAT): Only in participants where 10MWT is <12.5s at baseline
* Timed up and go test (TUG)
* Functional Ambulation Category (FAC)
* Health Related Quality of Life (HRQoL) via AQoL-4D

Description of intervention:

Control Group:

The control group will complete a suite of exercises based upon existing rehabilitation practices that aim to improve mobility after stroke. The supervising physiotherapist will select and progress the exercises, recording the performance of exercises in an exercise log and detailing incidence of adverse events. Exercise selection will include: gait retraining, cardiovascular fitness, lower limb strengthening, static and dynamic balance

Experimental group:

The experimental group will complete jump squats on the leg sled, single leg toe push offs (or bilateral where unable to complete single), alternating legs (i.e. bounding), mini tramp jumping, progressing to jogging, quick hip flexion and bounding on land.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at Caulfield Hospital Neurological Rehabilitation Unit at the time of recruitment
* Diagnosis of first stroke
* Presence of lower limb weakness determined by >10% difference in knee extensor strength between sides
* Functional Ambulation Category (FAC) > 3
* Can walk a minimal distance of 14 metres (to allow measurement on a 10metre walk test (10MWT)

Participants who meet all the inclusion criteria except for their FAC score will have their FAC score re-measured on a weekly basis until they reach a score of greater than or equal to 3, at which point they become eligible and will be approached for recruitment.

Exclusion Criteria:

* Unable to provide informed consent (determined by consultation with rehabilitation consultant and the team neuropsychologist)
* Other diagnosed central nervous system disorder affecting mobility
* Active oncological diagnosis
* Unstable medication condition such as unstable diabetes or unstable cardiac condition that would prevent participation in cardiovascular activity
* Recent orthopaedic trauma and/or osteoarthritis that would limit participation in physical exercise
* Not willing to continue to attend the program if they discharge home before the end of the six week program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 weeks
  Recruitment:
  * Number of stroke admissions to Caulfield Hospital
  * Number of stroke admissions that meet the inclusion/exclusion criteria
  * Number of those eligible who consent to participate
  Retention/Attrition:
  * Drop out rates over the six week period and reasons for drop outs
  * Number of sessions attended out of 18 over the six week period
  Clinical feasibility
  * Capacity of participants to perform the required exercises
  * Level of assistance required by therapist to perform the exercises - i.e. independent, supervision, assisted
  * Barriers to completing the required exercises during a session, i.e. incidence of delayed onset muscle soreness, fatigue
  * To be recorded for every session
  Safety
  * Incidence of adverse events
  * Types of adverse events
  * To be recorded for every session

SECONDARY OUTCOMES:
10 metre walk test comfortable pace | Baseline and 6 weeks
  Participants will be measured at comfortable gait speed. The middle 10metres of a 14 metre track will be recorded. The participant will be asked to walk at their own comfortable speed. There will be a cone at the start and finish of the 14metre track to guide participants and the middle 10 metres will be recorded.
10 metre walk test, maximum safe pace | Baseline and 6 weeks
  Same set-up as 10MWT comfortable pace, however the participant will be asked to walk as fast as they safely can without breaking into a run.
High level mobility assessment tool (HiMAT) | Baseline and 6 weeks
  The HiMAT is a 13 item assessment tool designed to assess high level walking tasks, the ability to negotiate stairs and the ability to run, hop, skip and jump. The HiMAT will be used to evaluate performance for higher level participants in the study where their 10MWT result may have a ceiling effect (where participants complete 10MWT in under 12.5seconds).
Timed up and go test (TUG) | Baseline and 6 weeks
  The TUG is highly reliable in stroke populations and correlates with walking performance and incidence of falls. Participants will be measured on the TUG from a 45cm chair. The will be asked to complete the test at their own comfortable speed.
Functional Ambulation Category (FAC) | Baseline and 6 weeks
  The FAC is a simple tool which uses an ordinal scale of 1 to 6 to measure the level of assistance a person requires to walk, and the different types of terrain they can manage such as indoors vs. outdoors, slopes and inclines.
Assessment of quality of life 4D | Baseline and 6 weeks
  Health related quality of Life will be measured using the Assessment of quality of life 4D. This has been shown to be a valid and sensitive measure in stroke, and has been used to determine the effects of mobility on HRQoL in neurological populations.

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve C Hendrey, B Phys (Hons), Principal Investigator — The Alfred; Anne E Holland, PhD, Principal Investigator — Alfred Health and La Trobe University; Gavin Williams, PhD, Principal Investigator — Epworth Healthcare, Melbourne University, La Trobe University; Ross Clark, PhD, Principal Investigator — Australian Catholic University
Locations (1):
- Alfred Health - Caulfield Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Hendrey G, Clark RA, Holland AE, Mentiplay BF, Davis C, Windfeld-Lund C, Raymond MJ, Williams G. Feasibility of Ballistic Strength Training in Subacute Stroke: A Randomized, Controlled, Assessor-Blinded Pilot Study. Arch Phys Med Rehabil. 2018 Dec;99(12):2430-2446. doi: 10.1016/j.apmr.2018.04.032. Epub 2018 May 30. PMID 29859180